CLINICAL TRIAL: NCT00180882
Title: LMBA02 Protocol for Patients With a Burkitt Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMBA02
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Burkitt Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Rituximab

INTERVENTIONS:
Drug: rituximab

SUMMARY:
To explore in a multicenter international prospective randomized study (phase III) whether rituximab combined with the standard French LMB chemotherapy scheme results in a higher rate of EFS than the LMB chemotherapy scheme alone in patients older than 18 years with Burkitt lymphoma or ALL 3.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18 years or older
* Histologically or cytologically proven Burkitt lymphoma according to the WHO classification
* WHO performance < 3
* Informed consent

Exclusion Criteria:

* Known HIV positive infection
* Positive serology for HCV and HBV (except after vaccination)
* Patients previously treated for lymphoma
* cardiac disease that contradict anthracycline chemotherapy
* Psychological or psychiatric condition who contradict steroids therapy
* Patients with serious renal failure unrelated to the lymphoma (serum creatinin level higher than 150 mmole/L)
* Cirrhosis or severe hepatic failure unrelated to the lymphoma
* Previous malignant disease except basal cell skin carcinoma or in situ uterine cervix carcinoma
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Primary organ transplant or other immunosuppressive conditions Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260
Dates: Start 2004-10

PRIMARY OUTCOMES:
Event free survival from date of first randomization

SECONDARY OUTCOMES:
Complete and partial response rate, overall survival, toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Vincent RIBRAG, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- [Derived] Ribrag V, Koscielny S, Bosq J, Leguay T, Casasnovas O, Fornecker LM, Recher C, Ghesquieres H, Morschhauser F, Girault S, Le Gouill S, Ojeda-Uribe M, Mariette C, Cornillon J, Cartron G, Verge V, Chassagne-Clement C, Dombret H, Coiffier B, Lamy T, Tilly H, Salles G. Rituximab and dose-dense chemotherapy for adults with Burkitt's lymphoma: a randomised, controlled, open-label, phase 3 trial. Lancet. 2016 Jun 11;387(10036):2402-11. doi: 10.1016/S0140-6736(15)01317-3. Epub 2016 Apr 11. PMID 27080498